CLINICAL TRIAL: NCT00046514
Title: A Phase II Clinical Trial of ABI-007 (A Cremophor-Free, Protein Stabilized, Nanoparticle Paclitaxel)Administered Weekly in Taxol Resistant Patients With Metastatic Breast Cancer
Brief Title: ABI-007 in Taxol Resistant Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA013
Record Dates: First submitted 2002-09-30; First posted 2002-10-03 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Breast Neoplasms; Metastases, Neoplasm
Keywords: Metastatic Breast Cancer; Taxol
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Albumin-Bound Paclitaxel

INTERVENTIONS:
Drug: ABI-007

SUMMARY:
The anticancer agent paclitaxel (marketed as Taxol) has shown remarkable activity against metastatic breast cancer. However, the Taxol formulation requires prolonged administration times, and there are safety problems that have been attributed to the solvent rather than the active ingredient, paclitaxel. This is a new formulation of paclitaxel that has been found to have fewer safety problems than Taxol, and may be administered safely at higher doses. This study will investigate the safety and efficacy of this new formulation of paclitaxel given intravenously once a week for three weeks, followed by a rest week. This cycle will be repeated until safety problems or treatment failure require that the patient stop therapy.

DETAILED DESCRIPTION:
The anticancer agent paclitaxel (Taxol for Injection Concentrate, Bristol-Meyers Squibb) has a broad spectrum of activity against several human cancers including carcinomas of ovary, breast, lung, esophagus and head and neck cancer. Taxol has shown remarkable activity against metastatic breast cancer, yielding response rates in the range of 40% to 60% in chemotherapy-naive patients and 25%-30% in patients refractory to anthracycline-containing regimens (Taxol package insert). The major limitation of Taxol is its poor water soluability requiring Cremophor (containing castor oil and ethanol) as a solvent. Taxol in this vehicle must be administered over 3-24 hours, and hypersensitivity reactions to Cremophor require a premedication routine of a corticosteroid, an antihistamine, and an H2 antagonist.

In this study, the test medication (ABI-007) is a nanoparticle colloidal composition of protein-stabilized paclitaxel that is reconstituted in saline. The infusion time for ABI-007 is minimal compared to Taxol (under an hour), and there is no premedication required. The maximally tolerated dose of this formulation of paclitaxel is 300 mg/m2, as compared to 175 mg/m2 for Taxol. As tumor response has been shown to be dose-dependent for paclitaxel, a higher dose allows for a potentially better response.

This open-label, Phase II study will determine the safety, tolerability and anti-tumor effect of ABI-007 monotherapy administered weekly in patients with metastatic breast cancer that have been previously treated with Taxol.

ELIGIBILITY:
Patients must be:

* If female, non-pregnant and not lactating, with a negative serum pregnancy test, and either not of child-bearing potential or practicing an approved contraception method
* Eighteen years of age or older
* Karnofsky Perfomance Status of 70% or 0-2 SWOG Performance Status
* No other malignancy, except non-melanoma skin cancer, CIN, or in-situ cervical cancer
* Measurable disease
* Suitable candidate for treatment with paclitaxel
* Previously treated with Taxol weekly or every three weeks, including adjuvant therapy, for metastatic breast cancer and relapsed within 12 months
* If, at baseline, patient has absolute neutrophil count of at least 1500 cells/mm3, platelet count of at least 100,000 cells/mm3,and hemoglobin of at least 9 g/dL
* If, at baseline, patient has AST and ALT of less than or equal to 2.5 x the upper limit of normal range; a total bilirubin less than or equal to 1.5 mg/dL; creatinine levels less than or equal to 2 mg/dL; and alkaline phosphatase levels less than or equal to 5 x the upper limit of normal range (unless there are bone but not liver metastases)
* Patient has an expected survival of at least 12 weeks
* Patient or his/her representative has signed an informed consent statement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2001-06

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Hawkins, M.D., Study Director — Celgene Corporation
Locations (1):
- Abraxis BioScience, Inc., Raleigh, North Carolina, United States

REFERENCES:
- [Background] Blum JL, Savin MA, Edelman G, Pippen JE, Robert NJ, Geister BV, Kirby RL, Clawson A, O'Shaughnessy JA. Phase II study of weekly albumin-bound paclitaxel for patients with metastatic breast cancer heavily pretreated with taxanes. Clin Breast Cancer. 2007 Dec;7(11):850-6. doi: 10.3816/CBC.2007.n.049. PMID 18269774